CLINICAL TRIAL: NCT04449406
Title: Early Detection of Pancreatic Adenocarcinoma (PDAC) Using a Panel of Biomarkers (UroPanc)
Brief Title: Early Detection of Pancreatic Adenocarcinoma (PDAC) Using a Panel of Biomarkers
Acronym: UroPanc
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: University of Liverpool (Other); University College, London (Other); Imperial College London (Other); Pancreatic Cancer Research Fund (Unknown); Ospedale San Raffaele (Other)
Responsible Party: Sponsor
Other Study IDs: 012335QM
Record Dates: First submitted 2020-05-05; First posted 2020-06-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Biomarker; PDAC; Pancreatic cancer; CA19-9; Urine
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine and blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals at risk of developing PDAC: * Symptomatic participants (via direct recruitment to UroPanc and via study/tissue bank(s) i.e. UCL ADEPTs study)
  * Asymptomatic participants (via study/tissue bank(s) i.e. University of Liverpool EUROPAC registry)
  Medical history, demographic information and concomitant medications information will be collected at baseline, together with blood and urine samples. Urinary biomarkers and plasma CA19-9 will be measured and the results compared with imaging data (and pathology, if it becomes available).

SUMMARY:
Urine and blood samples are being collected from patients with and without diseases of the pancreas. These samples will be tested with the aim of developing an accurate way of diagnosing diseases of the pancreas using the results.

DETAILED DESCRIPTION:
The main aim of this research study is to establish the accuracy of a urinary biomarker panel (LYVE1, REG1B, TFF1), and affiliated PancRISK score alone or in combination with plasma CA19-9 for early detection of pancreatic ductal adenocarcinoma (PDAC).

Samples will be collected from symptomatic individuals with suspected pancreatic cancer, and asymptomatic subjects at risk of developing PDAC.

The results of urine biomarker and CA19-9 analysis carried out on these samples will be compared to the imaging and, where available, histopathology data, which will inform the development of a predictive model to detect PDAC earlier.

ELIGIBILITY:
Inclusion criteria (Symptomatic patients):

* Able and willing to give informed consent
* ≥18 years old
* Suspected pancreatic diseases with symptoms including, but not limited to, diarrhoea, back pain, abdominal pain, nausea, vomiting, constipation or new onset diabetes

Exclusion criteria (Symptomatic patients):

* Current or prior treatment (chemotherapy, radiotherapy, surgical resection, biological therapy, and immunotherapy) for any malignancy other than basal cell carcinoma within 5 years of enrolment.

Asymptomatic participants will be identified through the EUROPAC registry and will fulfil EUROPAC's eligibility criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Samples from symptomatic and asymptomatic individuals at risk of PDAC will be provided to the UroPanc team by collaborating centres via dedicated tissue banks/registries already in place at UCL (ADEPTS) and the University of Liverpool (EUROPAC).
  Symptomatic individuals at risk which are being referred to specialist care by their general practitioners (GPs) will be recruited to participate in UroPanc when attending clinics (gastroenterology clinics, endoscopy units and Multidisciplinary Diagnostic Centres (MDCs)) at a participating study site.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of biomarker panel and affiliated risk score | Baseline until completion of standard-of-care diagnostic testing (up to 12 months after enrolment)
  Test accuracy, as measured by sensitivity/specificity (SN/SP) and positive predictive value/negative predictive value (PPV/NPV).

SECONDARY OUTCOMES:
Accuracy of biomarker panel and affiliated risk score when combined with CA19-9 result | Baseline until completion of standard-of-care diagnostic testing (up to 12 months after enrolment)
  Test accuracy, as measured by sensitivity/specificity (SN/SP) and positive predictive value/negative predictive value (PPV/NPV).
Economic and social impact of using biomarker panel for PDAC testing | Baseline until completion of standard-of-care diagnostic testing (up to 12 months after enrolment)
  Stakeholder and health economics analyses of the inclusion of the urine test into the existing diagnostic and surveillance pathways for PDAC.

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Crnogorac-Jurcevic, MD, PhD, Principal Investigator — Queen Mary University of London
Locations (4):
- United Kingdom (4):
  - EUROPAC study, University of Liverpool, Liverpool
  - ADEPTS study, University College London, London
  - Imperial College London, London
  - Royal London Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Radon TP, Massat NJ, Jones R, Alrawashdeh W, Dumartin L, Ennis D, Duffy SW, Kocher HM, Pereira SP, Guarner posthumous L, Murta-Nascimento C, Real FX, Malats N, Neoptolemos J, Costello E, Greenhalf W, Lemoine NR, Crnogorac-Jurcevic T. Identification of a Three-Biomarker Panel in Urine for Early Detection of Pancreatic Adenocarcinoma. Clin Cancer Res. 2015 Aug 1;21(15):3512-21. doi: 10.1158/1078-0432.CCR-14-2467. PMID 26240291
- [Background] Blyuss O, Zaikin A, Cherepanova V, Munblit D, Kiseleva EM, Prytomanova OM, Duffy SW, Crnogorac-Jurcevic T. Development of PancRISK, a urine biomarker-based risk score for stratified screening of pancreatic cancer patients. Br J Cancer. 2020 Mar;122(5):692-696. doi: 10.1038/s41416-019-0694-0. Epub 2019 Dec 20. PMID 31857725